CLINICAL TRIAL: NCT04803240
Title: Survey: Evaluation of Ocular Surface Disease Symptoms and Patient Satisfaction With Thealoz® Duo After 84 Days of Daily Treatment
Status: Completed | Type: Observational
Sponsor: Laboratoires Thea (Industry)
Collaborators: Iris Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: LT2280-PIV-0718
Record Dates: First submitted 2021-02-25; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Thealoz Duo — Non applicable
  Other Names: sodium hyaluronate and trehalose

SUMMARY:
Multi-centre, international, non-interventional, prospective survey

DETAILED DESCRIPTION:
To assess after 84 days, on a large scale patient population, the evaluation of ocular surface diseases and the satisfaction of dry eye disease (DED) treatment naïve patients or those who had to switch for tolerance, dissatisfaction or efficacy reasons to Thealoz® Duo.

ELIGIBILITY:
Inclusion Criteria:

* All dry eye patients who require artificial tears or need to change their current artificial tears for any reason (i.e. due to dissatisfaction or low efficacy, etc…)
* Outpatients of either sex, aged at least 18 years
* Patients informed of the objectives of the survey and agreeing to participate.

Exclusion Criteria:

* Use of cyclosporine, lifitegrast, tacrolimus, sirolimus within last 3 months and during the survey
* Use of topical ophthalmological treatments (glaucoma, etc…)
* Use of lacrimal plugs
* Ocular surgery in the last 12 months
* Concomitant use of corticosteroids
* Concomitant use of autologous serum or any blood derivatives
* Severe blepharitis
* Severe dry eye associated to

  * Eyelid malposition
  * Corneal dystrophy
  * Ocular neoplasia
  * Sjogren syndrome
  * Any systemic pathologies
* Pregnancy/lactation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All dry eye patients who require artificial tears or need to change their current artificial tears for any reason (i.e. due to dissatisfaction or low efficacy, etc…)
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
OSDI | 84 days
  Change from baseline for patient symptoms using the ocular surface disease index (OSDI©) questionnaire at Day 84. The OSDI is assessed on a scale of 0 to 100, with higher scores representing greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio MATEO, Dr., Principal Investigator — Hospital Miguel Servet; Philip BUCKHURST, Dr., Principal Investigator — University of Plymouth
Locations (1):
- University of Plymouth, Plymouth, United Kingdom

REFERENCES:
- [Derived] Mateo-Orobia AJ, Farrant S, Del-Prado-Sanz E, Blasco-Martinez A, Idoipe-Corta M, Lafuente-Ojeda N, Pablo-Julvez LE. A Preservative-Free Combination of Sodium Hyaluronate and Trehalose Improves Dry Eye Signs and Symptoms and Increases Patient Satisfaction in Real-Life Settings: The TEARS Study. Ophthalmol Ther. 2024 Dec;13(12):3123-3134. doi: 10.1007/s40123-024-01044-4. Epub 2024 Oct 21. PMID 39432158